CLINICAL TRIAL: NCT05547074
Title: Development and Validation of a New Prognostic Score Model Combining TNM Stage With Immune Risk Factors for Postoperative Pancreatic Ductal Adenocarcinoma
Brief Title: A New Prognostic Score Model for Pancreatic Ductal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Head of Hepatobiliary and Pancreatic Surgery, Zhejiang University
Other Study IDs: PSMPDAC
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Neoplasms Pancreatic
Keywords: pancreatic ductal adenocarcinoma; prognostic model; tumor-infiltrating immune cell; staging
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The training cohort: To develop the prognostic model, 302 cases of postoperative PDAC were included in the final analysis and divided into the training and validation cohort by stratified sampling with 7:3 ratio (The training cohort: n=212; The validation cohort: n=90).
  Interventions: Procedure: pancreatic cancer surgery
- The validation cohort: To develop the prognostic model, 302 cases of postoperative PDAC were included in the final analysis and divided into the training and validation cohort by stratified sampling with 7:3 ratio (The training cohort: n=212; The validation cohort: n=90).
  Interventions: Procedure: pancreatic cancer surgery

INTERVENTIONS:
Procedure: pancreatic cancer surgery — Surgical resection of pancreatic cancer，including radical or palliative surgery

SUMMARY:
The AJCC TNM staging system is the prevailing method in prognostic evaluation of pancreatic ductal adenocarcinoma (PDAC) at present , but it did not include factors such as the tumor immune microenvironment that are known to exert a profound impact on patients'clinical outcome. This study was aimed to develop a comprehensive and effective prognostic score model to predict prognosis and guide clinical management for postoperative PDAC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed PDAC
2. Achievement of surgical resection (including radical or palliative surgery)

Exclusion Criteria:

1. Lost to follow-up
2. Simultaneous presence of other tumors
3. Died in three months after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PDAC cases that underwent surgical resection (including radical or palliative surgery) from January 2016 to August 2019 were retrospectively reviewed and the survival follow-up (more than 14 months) was performed.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
overall survival | after pancreatic cancer surgery until october 31, 2020
  the number of months from the date of surgery to the date of the last follow-up visit or time of death.

SECONDARY OUTCOMES:
disease-free survival disease-free survival disease-free survival disease-free survival | after pancreatic cancer surgery until october 31, 2020
  the number of months from the date of surgery to the date of first confirmable recurrence or death

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Principal Investigator — First Affiliated Hospital, Medical College of Zhejiang University
Locations (1):
- First Affiliated Hospital, Medical College of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes